CLINICAL TRIAL: NCT04464733
Title: A Phase I Study to Evaluate the Safety, Tolerability and PK, PD of Oral HRS9950 in Healthy Subjects With Single or Multiple Dose and Chronic Hepatitis B Patients With Multiple Dose, and Food Effects of HRS9950 in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics(PK), Pharmacodynamics(PD) and Food Effect of HRS9950 in Healthy and CHB Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HRS9950-101
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (15):
- Treatment group A (Experimental): single dose
  Interventions: Drug: HRS9950; Drug: Placebo
- Treatment group B (Experimental): single dose
  Interventions: Drug: HRS9950; Drug: Placebo
- Treatment group C (Experimental): single dose; food effect
  Interventions: Drug: HRS9950; Drug: Placebo
- Treatment group D (Experimental): single dose
  Interventions: Drug: HRS9950; Drug: Placebo
- Treatment group E (Experimental): single dose
  Interventions: Drug: HRS9950; Drug: Placebo
- Treatment group F (Experimental): multiple doses
  Interventions: Drug: HRS9950; Drug: Placebo
- Treatment group G (Experimental): multiple doses
  Interventions: Drug: HRS9950; Drug: Placebo
- Treatment group H (Experimental): multiple doses
  Interventions: Drug: HRS9950; Drug: Placebo
- Treatment group I (Experimental): multiple doses
  Interventions: Drug: HRS9950; Drug: Placebo
- Treatment group J (Experimental): multiple doses
  Interventions: Drug: HRS9950; Drug: Placebo
- Treatment group K (Experimental): single dose
  Interventions: Drug: HRS9950; Drug: Placebo
- Treatment group L (Experimental): single dose
  Interventions: Drug: HRS9950; Drug: Placebo
- Treatment group M (Experimental): single dose
  Interventions: Drug: HRS9950; Drug: Placebo
- Treatment group N (Experimental): multiple doses
  Interventions: Drug: HRS9950; Drug: Placebo
- Treatment group O (Experimental): multiple doses
  Interventions: Drug: HRS9950; Drug: Placebo

INTERVENTIONS:
Drug: HRS9950 — HRS9950
Drug: Placebo — Placebo

SUMMARY:
The study is a randomized, Double-Blind, Placebo-Controlled study to evaluate the safety, tolerability and pharmacokinetics, pharmacodynamics and food effect of HRS9950. The study will be conducted in three parts sequentially:

Part 1, evaluate the safety, tolerability and pharmacokinetics, pharmacodynamics of single doses and multiple dose of HRS9950 tablet in healthy subjects. Part 1 will consist of 84 healthy subjects, 8 groups.There will be 14 subjects in 0.75mg dose group,10 subjects in each other dose group .

Part 2, evaluate food effect of HRS9950 in healthy subjects. Part 2 will consist of 14 healthy subjects, 1 group (one of groups in Part 1).

Part 3, evaluate the safety, tolerability and pharmacokinetics, pharmacodynamics of multiple doses of HRS9950 tablet in naive and treatment-experienced chronic hepatitis B (CHB) patients. Part 3 will consist of 60 CHB patients, 1 group for naive patients and 5 groups for treatment-experienced patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

  1. Signed informed consent.
  2. Aged 18~55.
  3. Body weight ≥ 50 kg for male; ≥ 45 kg for female, body mass index (BMI) between 18 to 28 kg/m2.
  4. Vital signs, physical examination, laboratory results are within normal range or considered not clinically significant.
  5. Female subjects (including partner) of childbearing potential must be using a medically acceptable form of birth control.
* CHB subjects

  1. Signed informed consent.
  2. Aged 18~65.
  3. CHB subjects should meet the following two criteria:

  <!-- -->

  1. IgM HBcAb negative and HBsAg positive.
  2. Two recorded HBsAg positive, and the time interval between the two tests was at least 6 months, one of which was the result of this screening 4. Treatment-experienced CHB subjects should also meet the following criteria:

  <!-- -->

  1. Have received nucleoside analogue treatment for at least 6 months
  2. HBeAg positive or negative, and the HBV DNA concentration should be less than 20 IU/mL for at least 6 months before enrollment
  3. Confirm ALT <1.5 ULN (upper limit of normal value) by two measurements within 6 months before enrollment 5. Treatment-naïve CHB subjects should also meet the following criteria:

  <!-- -->

  1. Have not received antiviral therapy (nucleosides or interferons) at screening
  2. HBeAg positive or negative, and the HBV DNA concentration should be greater than 2000 IU/mL for at least 6 months before enrollment
  3. Confirm ALT> 1 ULN by two measurements within 6 months before enrollment 6. Female subjects (including partner) of childbearing potential must be using a medically acceptable form of birth control.

Exclusion Criteria:

* Healthy subjects

  1. Currently suffering from cardiovascular, liver, kidney, digestive, nervous, blood, thyroid or mental diseases.
  2. Medical history of malignant tumor.
  3. Have a digestive system disease or a medical history of severe digestive system disease.
  4. Have severe infection, severe trauma or major surgical operations within 3 months.
  5. 12-ECG test have clinical significant abnormality or the QT interval (QTc) > 450 ms.
  6. Clinical laboratory examinations or chest radiographs have clinical significant abnormality.
  7. Have a medical history of immune-mediated diseases.
  8. Screening for infectious diseases is positive (Including HBsAg, Anti-HCV, TPPA, Anti-HIV).
  9. Suspected allergy to any ingredient in the study drug.
  10. Have any drug that inhibits or induces liver metabolism within 1 month.
  11. Take any prescription drugs, over-the-counter drugs and Chinese herbal medicines within 14 days before taking the study drug, or took any drugs within 5 half-lives at the time of screening; plan to take other drugs during the test period.
  12. Participated in clinical trials of any drug or medical device within 3 months before screening, or within 5 half-lives before screening.
  13. Had donated blood or blood transfusion in 8 weeks or ≥ 400 mL within 3 months prior to screening or ≥ 200 mL within 1 months.
  14. The average daily smoking ≥ 5 cigarettes within three months; the average daily alcohol intake in a month exceeds 15 g (15 g alcohol is equivalent to 450 mL beer or 150 mL wine or 50 mL low-alcohol);
  15. Keep smoking, drinking alcohol or consuming caffeinated foods or beverages (more than 8 cups, 1 cup = 250 mL) 2 days before taking the study drug and during the study; and those who have special dietary requirements and cannot follow the unified diet;
  16. Pregnant or lactating women;
  17. Drug screening or alcohol breath test is positive.
  18. Other conditions that the investigator believes the subject is not suitable.
* CHB subjects

  1. Currently suffering from serious cardiovascular, liver, kidney, digestive, nervous, blood, thyroid or mental diseases other than hepatitis B.
  2. People have acute or chronic liver disease by non-HBV infection.
  3. Liver stiffness (LSM)> 12.4 kPa by noninvasive transient liver elastography (eg Fibroscan®) or recorded liver biopsy suggesting cirrhosis or extensive fibrosis
  4. Primary liver cancer, high-risk groups of primary liver cancer or AFP> 50g/L;
  5. Have clinically demonstrated or history of liver function decompensation, including but not limited to: hepatic encephalopathy, hepatorenal syndrome, splenomegaly, ascites, etc.;
  6. Laboratory inspection:

     1. Platelet count <90×109/L;
     2. White blood cell count <3.0×109/L;
     3. Absolute value of neutrophils <1.5×109/L;
     4. Serum total bilirubin>2×ULN;
     5. Albumin <30 g/L;
     6. Creatinine clearance rate ≤60ml/min;
     7. INR>1.5;
     8. ALT exceeds 5 times the upper limit of normal value on screening/baseline visit
  7. HIV and/or syphilis antibody positive
  8. Subjects who have previously received organ/bone marrow transplantation;
  9. Have used immunosuppressants, immunomodulators or cytotoxic drugs within 6 months before the study medication;
  10. Suspected allergy to any ingredient in the study drug.
  11. The average daily smoking ≥ 5 cigarettes within three months; the average daily alcohol intake in a month exceeds 15 g (15 g alcohol is equivalent to 450 mL beer or 150 mL wine or 50 mL low-alcohol);
  12. Keep smoking, drinking alcohol or consuming caffeinated foods or beverages (more than 8 cups, 1 cup = 250 mL) 2 days before taking the study drug and during the study; and those who have special dietary requirements and cannot follow the unified diet;
  13. Pregnant or lactating women;
  14. Drug screening or alcohol breath test is positive.
  15. Other conditions that the investigator believes the subject is not suitable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of treatment-related adverse events as assessed by CTCAE v5.0 | 8 DAYS for Group A-M; 29 DAYS for Group F; 50 DAYS for Group G-O
Maximum Plasma Concentration [Cmax] | 0-48 hours after each dose for Group A-E、K-M；Group F- J、N、O at Day 1 and Day 22
  Pharmacokinetic parameters of HRS9950, main metabolite and identified major metabolites in plasma
Area under the concentration time curve [AUC] | 0-48 hours after each dose for Group A-E、K-M；Group F- J、N、O at Day 1 and Day 22
  Pharmacokinetic parameters of HRS9950, main metabolite and identified major metabolites in plasma
Time to maximum plasma concentration [Tmax] | 0-48 hours after each dose for Group A-E、K-M；Group F- J、N、O at Day 1 and Day 22
  Pharmacokinetic parameters of HRS9950, main metabolite and identified major metabolites in plasma
Apparent clearance [CL/F] | 0-48 hours after each dose for Group A-E、K-M；Group F- J、N、O at Day 22
  Pharmacokinetic parameters of HRS9950, main metabolite and identified major metabolites in plasma
Half-time [t1/2] | 0-48 hours after each dose for Group A-E、K-M；Group F- J、N、O at Day 22
  Pharmacokinetic parameters of HRS9950, main metabolite and identified major metabolites in plasma
Apparent volume of distribution [Vz/F（Vd）] | 0-48 hours after each dose for Group A-E、K-M；Group F- J、N、O at Day 22
  Pharmacokinetic parameters of HRS9950, main metabolite and identified major metabolites in plasma
Mean residence time [MRT] | 0-48 hours after each dose for Group A-E、K-M；Group F- J、N、O at Day 22
  Pharmacokinetic parameters of HRS9950, main metabolite and identified major metabolites in plasma
The concentration of IL-12p40 in the serum | 0-48 hours after each dose for Group A-E、G-O
  After single or multiple administration of HRS9950

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Youan Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided